CLINICAL TRIAL: NCT02086084
Title: Extra-corporeal CO2 Removal as an Adjunct to Non-Invasive Ventilation in Acute Severe Exacerbations of COPD
Brief Title: ECCO2R as an Adjunct to NIV in AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Alung Technologies (Industry)
Responsible Party: Principal Investigator, Nicholas Barrett, Consultant in Critical Care, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECCO2R in AECOPD
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute Exacerbation Chronic Obstructive Pulmonary Disease; AECOPD; Non invasive ventilation; NIV; Extracorporeal carbon dioxide removal; ECCO2R
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV (Active Comparator): Standard application of NIV in hypercapnic respiratory failure as per usual standard of care
  Interventions: Device: NIV
- ECCO2R (Experimental): Addition of ECCO2R to NIV in AECOPD
  Interventions: Device: NIV; Device: ECCO2R

INTERVENTIONS:
Device: NIV — Standard care
Device: ECCO2R — Application of ECCO2R in addition to NIV
  Other Names: Haemolung
  Arms: ECCO2R

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the UKs commonest chronic diseases and is responsible for a significant number of acute hospital admissions. COPD is characterised by progressive destruction in the elastic tissue within the lung, causing respiratory failure. The clinical course of COPD is characterised by recurrent acute exacerbations (AECOPD), causing considerable morbidity and mortality. Patients with moderate to severe acute exacerbations present with increased work of breathing and hypercapnia. The standard for respiratory support in this setting is non-invasive ventilation (NIV), a management strategy underpinned by a considerable evidence base. However despite NIV, up to 30% of patients with AECOPD will 'fail' and require intubation and mechanical ventilation. The mortality rate for patients requiring NIV is approximately 4%, if conversion to mechanical ventilation occurs the mortality is 29%.

The last decade has seen an increasing interest in the provision of extracorporeal support for respiratory failure. The key element that has underpinned improving survival has been technological advancement. This has resulted in pumps causing less blood trauma and inflammatory response, better percutaneous cannulation techniques and coated circuits with reduced heparin requirements. Overall this has significantly reduced the complications associated with the provision of extracorporeal support. One variation of this technique (extra-corporeal CO2 removal ECCO2R) allows CO2 clearance from the blood. This approach has been the subject of a number of animal experiments and uncontrolled human case series demonstrating improved arterial CO2 and reduced work of breathing. Our own unpublished series demonstrates the same physiological changes. However to date the benefits of this approach have not been tested in a randomised controlled trial.

The hypothesis is that the addition of ECCO2R to NIV will shorten the duration of NIV and reduce likelihood of intubation.

ELIGIBILITY:
Inclusion criteria

* Known COPD with an acute exacerbation. An acute exacerbation is defined as per the GOLD criteria as an increase in dyspnoea, cough and/or sputum over the patient's normal symptoms. A severe exacerbation is defined as one requiring hospital admission.
* Patients with a persistent arterial pH<7.30 due primarily to hypercapnic respiratory failure after standard medical therapy and at least 1 hour of NIV.
* Age over 18

Exclusion Criteria

* Haemodynamic instability after ensuring euvolaemia
* Acute multiple organ failure requiring other organ supportive therapy, including indication for intubation and mechanical ventilation
* Known allergy/intolerance of heparin including known heparin induced thrombosis and thrombocytopaenia
* Acute uncontrolled haemorrhage
* Intracerebral haemorrhage
* Recent (<6 months) ischaemic cerebrovascular accident
* Organ transplant recipient
* Expected to die within 24 hours
* Venous abnormality or body habitus precluding cannulation
* Contraindication to NIV (as per British Thoracic Society recommendation)

  * Facial burns/trauma/recent facial or upper airway surgery
  * Vomiting
  * Fixed upper airway obstruction
  * Undrained pneumothorax
  * Recent upper gastrointestinal surgery
  * Inability to protect the airway
  * Life threatening hypoxaemia (PaO2/FiO2 <20kPa)
  * Bowel obstruction
  * Patient refusal
* Pregnancy
* Severe hepatic failure (ascites, hepatic encephalopathy or bilirubin >100umol/L)
* Severe chronic cardiac failure (NYHA class III or IV)
* Bleeding diathesis (INR>1.5, platelets <80,000) in the absence of anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Time to cessation NIV | participants will be followed for the duration of ICU stay, an expected average of 4 days
  Time to cessation of NIV is defined as from NIV commencement to 6 hours without NIV.

SECONDARY OUTCOMES:
Mortality | at 90 days
Time to event analysis | initial phase of study, an expected average of 3 hours
  This is a composite endpoint to assess the ability to complete the required elements of the study from screening to commencement of ECCO2R in a clinically relevant timeframe
Health-related quality of life (HRQoL) | 90 days
Cannulation-related outcomes | participants will be followed for the duration of ICU stay, an expected average of 4 days
  composite outcome of cannulation related complications
haemolysis related to the intervention | participants will be followed for the duration of ICU stay, an expected average of 4 days
work of breathing | participants will be followed for the duration of ICU stay, an expected average of 4 days
Time to cessation ECCO2R | participants will be followed for the duration of ICU stay, an expected average of 4 days
  Defined as from the commencement of ECCO2R to 6 hours following cessation of CO2 removal
Time to normalisation of pH | participants will be followed for the duration of ICU stay, an expected average of 4 days
Hospital Length of stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
Intubation rate | participants will be followed for the duration of ICU stay, an expected average of 4 days
Incidence of tracheostomy | participants will be followed for the duration of ICU stay, an expected average of 4 days
length of ICU stay | participants will be followed for the duration of ICU stay, an expected average of 4 days
Tolerance of therapy | participants will be followed for the duration of ICU stay, an expected average of 4 days
subjective dyspnoea | participants will be followed for the duration of ICU stay, an expected average of 4 days
nutrition | participants will be followed for the duration of ICU stay, an expected average of 4 days
  total caloric intake during interventional period
Mobilisation | participants will be followed for the duration of ICU stay, an expected average of 4 days
  mobilisation from bed during the study period
thrombotic complications | participants will be followed for the duration of ICU stay, an expected average of 4 days
  measurement of thrombotic complications in the patient related to the device
respiratory mechanics | participants will be followed for the duration of ICU stay, an expected average of 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Barrett, FCICM, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Luigi Camporota, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Nicholas Hart, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Barrett NA, Murgolo F, Grasso S, Kostakou E, Hart N, Murphy P, Douiri A, Camporota L. Physiological Assessment of ECCO2R on the Work of Breathing in Exacerbations of COPD. COPD. 2024 Dec;21(1):2436169. doi: 10.1080/15412555.2024.2436169. Epub 2024 Dec 5. PMID 39639560
- [Derived] Barrett NA, Hart N, Daly KJR, Marotti M, Kostakou E, Carlin C, Lua S, Singh S, Bentley A, Douiri A, Camporota L. A randomised controlled trial of non-invasive ventilation compared with extracorporeal carbon dioxide removal for acute hypercapnic exacerbations of chronic obstructive pulmonary disease. Ann Intensive Care. 2022 Apr 21;12(1):36. doi: 10.1186/s13613-022-01006-8. PMID 35445986
- [Derived] Barrett NA, Hart N, Camporota L. In vivo carbon dioxide clearance of a low-flow extracorporeal carbon dioxide removal circuit in patients with acute exacerbations of chronic obstructive pulmonary disease. Perfusion. 2020 Jul;35(5):436-441. doi: 10.1177/0267659119896531. Epub 2020 Jan 11. PMID 31928313
- [Derived] Barrett NA, Kostakou E, Hart N, Douiri A, Camporota L. Extracorporeal carbon dioxide removal for acute hypercapnic exacerbations of chronic obstructive pulmonary disease: study protocol for a randomised controlled trial. Trials. 2019 Jul 30;20(1):465. doi: 10.1186/s13063-019-3548-4. PMID 31362776